CLINICAL TRIAL: NCT04552223
Title: A Phase 2 Study of Nivolumab + BMS-986016 (Relatlimab) in Patients With Metastatic Uveal Melanoma
Brief Title: Nivolumab Plus Relatlimab in Patients With Metastatic Uveal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jose Lutzky, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jose Lutzky, MD, Director, Cutaneous Malignancies, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200847; CA224-094 (Other: Bristol-Myers Squibb); NCI-2020-11454 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Uveal Melanoma
Keywords: Metastatic Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab Plus Relatlimab Group (Experimental): Participants in this group will receive Nivolumab and Relatlimab administered together on Day 1 of every 4 week cycle. Both drugs will be administered until disease progression or intolerable toxicity for up to 24 months.
  Interventions: Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 480mg administered intravenously on Day 1 of each 4 week cycle.
  Other Names: Opdivo
Drug: Relatlimab — Relatlimab 160 mg administered intravenously on Day 1 of each 4 week cycle.
  Other Names: BMS-986016

SUMMARY:
The purpose of this research is to test if a combination treatment of nivolumab and relatlimab will result in tumor reduction in patients with metastatic uveal melanoma.

DETAILED DESCRIPTION:
This is a phase II single-institution trial with a Simon two-stage minimax design with 27 patients (13 in stage 1, 14 in stage 2) setting a 5% type I error and 80% power under true objective response rate (ORR) of 20%. The null hypothesis (ORR=5%) is rejected if 4 or more responses are observed in 27 patients. No prior PD-1, CTLA-4 and/or LAG-3 blocking antibody treatment was allowed. We will also perform single-cell mRNA and T-cell receptor (TCR) variable, diversity, and joining (V[D]J) sequencing pre-treatment and at either progression or response.

Patients will be treated with nivolumab 480 mg/relatlimab 160 mg IV q4wks to progression or intolerable toxicity for up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. Have a biopsy-proven diagnosis of metastatic uveal melanoma, previously untreated with anti-PD-1,Cytotoxic T lymphocyte antigen 4 (CTLA-4) and/or lymphocyte activation gene 3 (LAG-3) blocking antibodies.
2. Agree to undergo a pre-treatment and a post-treatment fresh biopsy of the tumor, if easily accessible and low-risk.
3. Have completed all previous therapy for a minimum of 3 weeks before the first dose of experimental treatment. All adverse events of previous therapy must have resolved. Palliative radiation therapy to a limited field is allowed within this 3 week period.
4. Be willing and able to provide written informed consent/assent for the trial.
5. Be ≥ 18 years of age on day of signing informed consent.
6. Have measurable disease based on RECIST 1.1.
7. Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
8. Left Ventricular Ejection Fraction (LVEF) assessment with documented LVEF 50% by either TTE or Multiple Gated Acquisition (MUGA) (TTE preferred test) within 6 months from first study drug administration
9. Demonstrate adequate organ function as defined in Table 1. All screening labs should be performed within 10 days of treatment initiation:

   * Hematological:

     * Absolute neutrophil count (ANC) ≥1,500 /microliter (mcL)
     * Platelets ≥100,000 / mcL
     * Hemoglobin ≥ 9 g/dL or ≥5.6 mmol/L (within 7 days of assessment)
   * Renal:

     * Serum creatinine ≤ 1.5 X upper limit of normal (ULN) OR
     * Measured or calculated a creatinine clearance ≥30 mL/min for subject with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl)
   * Hepatic:

     * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
     * Aspartate Aminotransferase (AST) (SGOT) and Alanine Amino Transferase (ALT) (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
     * Albumin ≥ 2.5 mg/dL
   * Coagulation:

     * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
     * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
     * Creatinine clearance should be calculated per institutional standard.
10. If a female of childbearing potential, have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. If a female of childbearing potential, be willing to use an adequate method of contraception as outlined in Section 5.8 Contraception, for the course of the study through 24 weeks after the last dose of study medication. Must abstain from ova donation for a minimum of 5 months after the end of treatment.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. If a male of childbearing potential, agree to use an adequate method of contraception as outlined in Section 5.8- Contraception, starting with the first dose of study therapy through 7 months after the last dose of study therapy. Must abstain from sperm donation for a minimum of 24 weeks after the end of treatment.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

1. Are currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of the first dose of treatment.
2. Have a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients on replacement doses of corticosteroids and patients who received steroids as pre-medication to prevent an imaging contrast allergy are allowed.
3. Have a known history of active tuberculosis (Bacillus Tuberculosis)
4. Have had prior treatment with a PD-1 and/or LAG-3 targeted agent
5. Have hypersensitivity to nivolumab, relatlimab or any of their excipients.
6. Have had a prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from clinically significant adverse events due to agents administered more than 3 weeks earlier.
7. Have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 3 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from clinically significant adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
   * Note: Patients will be allowed necessary and palliative radiation therapy to limited fields during the trial, as long as it does not encompass a target lesion.
8. Have a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma or squamous cell carcinoma of the skin that has undergone potentially curative therapy, in situ cervical cancer, ductal carcinoma in situ (DCIS), incidentally discovered asymptomatic thyroid cancer, Prostate Specific Antigen (PSA) recurrence of prostate cancer stable on hormonal therapy with no otherwise detectable disease, and a previous diagnosis of malignancy that has shown no evidence of disease progression for 5 years or longer.
9. Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis as well as a history of previous or current significant brain hemorrhage. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids to treat edema for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which will be excluded regardless of clinical stability.
10. Have active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Have known history of, or any evidence of active, non-infectious pneumonitis.
12. Have an active infection requiring systemic therapy.
13. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Have a diagnosis or known history of Human Immunodeficiency Virus (HIV), unless controlled on antiretroviral drugs and have undetectable levels of HIV antibodies.
17. Have known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C.
18. Have received a live vaccine within 30 days of planned start of study therapy.
19. Have a history of myocarditis, regardless of etiology
20. Have a troponin T (TnT) or I (TnI)

    * i) > 2x institutional upper limit of normal (ULN) : patient is excluded.
    * ii) between > 1 to 2 x ULN enrollment will be permitted if a repeat assessment remains < 2 x ULN and participant undergoes a cardiac evaluation and is cleared by a cardiologist or cardio-oncologist
21. Are patients with impaired decision-making capacity
22. Are prisoners or participants who are involuntarily incarcerated. (Note: under certain specific circumstances a person who has been imprisoned may be included as a participant. Strict conditions apply and Bristol-Myers Squibb approval is required).
23. Are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
24. Have psychological, familial, sociological, or geographical conditions that potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the participant before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2026-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Lutzky, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab Plus Relatlimab Group
Started | 27
Completed | 26
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab Plus Relatlimab Group
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) will be the percentage of study participants with a confirmed complete response (CR) or partial response PR to study therapy as per treating physician evaluation using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Up to 24 months
Population: Participants that completed at least two cycles of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab Plus Relatlimab Group
Number analyzed (Participants) | 26
percentage of participants | 7.7 [1 to 25.1]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) is the proportion of patients with confirmed complete response (CR), partial response (PR), or stable disease (SD) as per treating physician evaluation using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Up to 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from the date of enrollment to the date that objective progression disease is documented or death due to any cause, whichever occurs first.
Time Frame: Up to 4 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the date of enrollment to the date of death.
Time Frame: Up to 4 years
Reporting Status: Not Posted

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the time from the date of first documented response (CR or PR) until date of documented progression or death in the absence of disease progression.
Time Frame: Up to 4 years
Reporting Status: Not Posted

6. Secondary Outcome: Proportion of Study Participants With Treatment-Related Toxicity
Description: The safety profile of the study therapy will be determined by the proportion of study participants experiencing treatment-related adverse events (AEs) and serious adverse events (SAEs). AEs and SAEs will be tabulated by type, grade, severity, treatment attribution according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 25 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Nivolumab Plus Relatlimab Group
All-Cause Mortality (participants affected / at risk) | 17/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab Plus Relatlimab Group (N=27)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab Plus Relatlimab Group (N=27)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 13 (32)
Alkaline phosphatase increased (Investigations) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 13 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 9 (10)
Cardiac troponin T increased (Investigations) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Dizziness (Nervous system disorders) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dysuria (Renal and urinary disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Fatigue (General disorders) | 15 (23)
Fever (General disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 7 (7)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lipase increased (Investigations) | 5 (9)
Lymphocyte count decreased (Investigations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (8)
Nausea (Gastrointestinal disorders) | 8 (8)
Neutrophil count decreased (Investigations) | 1 (1)
Pain (General disorders) | 1 (2)
Papulopustular rash (Infections and infestations) | 1 (1)
Periorbital edema (Eye disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Pregnancy
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — COVID-19 positive
Serum amylase increased (Investigations) | 4 (7)
Sinusitis (Infections and infestations) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Thyroid stimulating hormone increased (Investigations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT04552223/Prot_SAP_000.pdf